CLINICAL TRIAL: NCT03993730
Title: Cardiovascular Magnetic Resonance GUIDEd Insertion of Implantable Cardiac Defibrillator in Dilated CardioMyopathy
Acronym: CMR GUIDE DCM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Flinders University (Other)
Responsible Party: Principal Investigator, Joseph Selvanayagam, Principal Investigator, Flinders University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CMRG-2
Record Dates: First submitted 2019-05-03; First posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Dilated Cardiomyopathy; Left Ventricular Systolic Dysfunction; Fibrosis Myocardial
MeSH Terms: conditions — Cardiomyopathy, Dilated; Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device Implantation (Other): A prospective, blocked, randomised, controlled trial of primary prophylaxis ICD therapy or ILR insertion in patients with LVEF <45% and LGE on CMR.
  Interventions: Device: ICD; Device: ILR
- Observational Registry (No Intervention): A prospective observational registry of patients with LVEF <45% and no LGE on CMR.

INTERVENTIONS:
Device: ICD — Insertion of ICD in patients with LVEF <45% and LGE on CMR.
  Arms: Device Implantation
Device: ILR — Insertion of ILR in patients with LVEF <45% and LGE on CMR.
  Arms: Device Implantation

SUMMARY:
CMR GUIDE DCM is a randomized controlled trial with a registry for non-randomized patients.

Patients enrolled will have non-ischemic cardiomyopathy (NICM) with mild to severe Left Ventricular (LV) systolic dysfunction with replacement fibrosis identified on Cardiac Magnetic Resonance (CMR).

954 patients will be randomised from 50 sites across 4-6 countries worldwide to receive an implantable defibrillator (ICD) or implantable loop recorder (ILR).

Device and clinical follow-up will be performed at 3, 6, 12, 24, 36 months and at end of study.

DETAILED DESCRIPTION:
The planned research will have two components: A prospective, blocked, randomized, controlled trial of primary prophylaxis ICD therapy or ILR insertion in patients with LVEF <45% and Late Gadolinium Enhancement (LGE) on CMR and

A prospective observational registry of patients with LVEF <45% and no LGE on CMR. Registry patients will not have an intervention but will have the same follow up frequency as the randomized patients.

The Primary objective is to determine if routine CMR guided management strategy of implantable defibrillator (ICD) insertion reduces total mortality compared to a conservative strategy of implantable loop recorder (ILR) insertion and standard care.

The secondary objectives include:

* To determine if routine CMR guided management strategy of ICD insertion reduces sudden cardiac death (SCD) compared to a conservative strategy of ILR insertion and standard care.
* To ascertain the rate of SCD in patients with DCM and LGE scar across a wide range of left ventricular ejection fraction (LVEF).

Statistical analysis will be performed on an intention-to-treat basis. The main analysis of time to death from any cause will be performed using a log- rank test.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than/equal to 18 years old
* Non-ischemic cardiomyopathy of dilated type
* Left Ventricular Ejection Fraction < 45%
* Able and willing to comply with all pre, post and follow-up testing and requirements
* On maximum tolerated doses of angiotensin converting enzyme (ACE) inhibitors (or Angiotensin Receptor Blockers(ARB) or Neprilysin Inhibitors) and Beta Blockers

Exclusion Criteria:

1. Known coronary artery disease (CAD) (History of Myocardial Infarction or Significant Epicardial CAD on Angiography)
2. Hypertrophic Cardiomyopathy
3. Cardiomyopathy related to sarcoidosis
4. Arrhythmogenic Right Ventricular Dysplasia
5. Standard LGE CMR contraindications (e.g. severe claustrophobia, metal)
6. Currently implanted permanent pacemaker and/or pacemaker/ICD lead
7. Clinical indication for ICD or pacemaker or Cardiac Resynchronisation Therapy
8. Contraindications to intravenous Gadolinium
9. Severe renal insufficiency (eGFR< 45mls/min/1.73m2 )
10. New York Heart Association Heart Failure functional class IV
11. Conditions associated with life expectancy <1 year
12. Pregnancy or in females of child-bearing potential, the non-use of accepted forms of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1880 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality | Through to study completion, an average of 4 years

SECONDARY OUTCOMES:
Number of Participants who have Sudden Cardiac Death | Through to study completion, an average of 4 years
Number of Participants who have a Haemodynamically significant ventricular arrhythmia event | Through to study completion, an average of 4 years
Quality of life assessed by Kansas City Cardiomyopathy Questionnaire | Measured at 3, 6, 12, 24, 36 months through to study completion
  The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. An overall summary score can be derived from the above 23 items which will be between 0-100. A higher score reflects a better health status.
Number of Participants who have a Heart Failure related hospitalisation | Through to study completion, an average of 4 years
Health economic evaluation of cost | At study completion, an average of 4 years
  Various different country jurisdictions will be chosen

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B Selvanayagam, MBBS, Principal Investigator — Flinders Medical Centre

IPD SHARING:
Plan to Share IPD: No